CLINICAL TRIAL: NCT05412433
Title: Clinic-based HIV Identification and Prevention Project Using Electronic Resources
Acronym: CHIPPER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Michigan (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: IRB00331706; 1R01MH132146 (NIH)
Record Dates: First submitted 2022-06-02; First posted 2022-06-09 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: HIV Prevention; Primary Care; PrEP
Keywords: HIV prevention; PrEP; Cis-gender women
MeSH Terms: interventions — Multilevel Analysis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (Active Comparator): Participants in this arm will receive standard of care
  Interventions: Behavioral: Control
- Patient Level + Multilevel (Experimental): Participants in the arm will receive the patient level and multi-level intervention
  Interventions: Behavioral: Patient Level; Behavioral: Multilevel
- Multilevel (Experimental): Participants in this arm will receive the multi-level intervention
  Interventions: Behavioral: Multilevel

INTERVENTIONS:
Behavioral: Patient Level — Electronic data collection with scoring, patient awareness of HIV risk score, patient viewing of PrEP animations
  Arms: Patient Level + Multilevel
Behavioral: Multilevel — Electronic data collection with scoring, patient awareness of HIV risk score, patient viewing of PrEP animations, provider electronic health records (EHR) alerts
  Arms: Multilevel; Patient Level + Multilevel
Behavioral: Control — Standard of care
  Arms: Standard of Care

SUMMARY:
Hybrid Type II effectiveness-implementation trial to investigate whether electronic medical and sexual history data collection with HIV risk categorization/scoring will increase pre-exposure prophylaxis (PrEP) uptake among cis-gender women attending routine well-woman gynecologic preventative visits.

DETAILED DESCRIPTION:
Forty-two Obgyn providers will be randomized into 1 of three arms. Patients of enrolled providers who attend an ObGyn clinic for any preventative visit will complete an electronic history form (eHxForm) before clinic through a message sent through the patient portal (MyChart), email, or secure text messaging. The sexual history questions will be scored and categorized into 3 categories. Patients with a low score (0-3) will receive an electronic message offering a laboratory HIV test per USPSTF guidelines. If she accepts, then an automated Epic order will be placed for the provider to sign during the office visit.

Patients with a medium/high score (4-10) will be assigned a study arm based on their provider's group (arm 1: control, arm 2: patient will view score and a PrEP video, arm 3: procedures in arm 2 PLUS providers will receive an electronic health record alert that the patient may have HIV risk factors. This will occur automatically via programming integrated into the electronic health record. The primary outcome is PrEP uptake. The implementation strategy will be evaluated using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework.

ELIGIBILITY:
Inclusion Criteria:

* Patients of enrolled providers aged 15-65 years
* Presenting for preventive care (i.e., well-woman exam, sexually transmitted infection testing, pre-conception counseling, or birth control).

Exclusion Criteria:

* Pregnant and has established prenatal care, i.e., visit is for prenatal care
* Non-English or non-Spanish speaking
* Living with HIV
* Unable to complete the eHxForm

Ages: 15 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Cisgender
Enrollment: 1170 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of PrEP prescriptions written for each patient | 4 weeks
  Number of PrEP prescriptions written for each patient up to 4 weeks after office visit.

SECONDARY OUTCOMES:
Cost-Effectiveness Analysis (Incremental cost-effectiveness ratios) | Approximately 5 years
  Incremental cost-effectiveness ratios
Cost-Effectiveness Analysis (Return on Investment) | Approximately 5 years
  Return on investment (intervention benefits, avoided direct medical costs, and incremental implementation costs)
Cost-Effectiveness Analysis (Total Budget) | Approximately 5 years
  Total budget to finance each intervention strategy (intervention and implementation costs)
Proportion of patients who complete the Electronic History Form (eHxForm) | 6 months
  Adoption of Electronic History Form as assessed by the proportion of consecutive eligible patients in each clinic who completed the eHxForm.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Powell, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Health System, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Izadi LH, Mmeje O, Drabo EF, Perin J, Martin S, Coleman JS. An effectiveness-implementation trial protocol to evaluate PrEP initiation among U.S. cisgender women using eHealth tools vs. standard care. Front Reprod Health. 2023 Jun 8;5:1196392. doi: 10.3389/frph.2023.1196392. eCollection 2023. PMID 37361343